CLINICAL TRIAL: NCT06894303
Title: Evaluation of Remote Programming of Cochlear Implants in Routine Cochlear Implant Follow-up
Status: Recruiting | Type: Observational
Sponsor: Advanced Bionics AG (Industry)
Responsible Party: Sponsor
Other Study IDs: ABInt-24-23
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Cochlear Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: Unilateral users
  Interventions: Device: Target CI v1.5 remote programming
- Group 2: Bilateral users
  Interventions: Device: Target CI v1.5 remote programming
- Group 3: Bimodal users
  Interventions: Device: Target CI v1.5 remote programming

INTERVENTIONS:
Device: Target CI v1.5 remote programming — Use of the remote programming function of Target CI v1.5 and the AB remote support application

SUMMARY:
This is a prospective and monocentric clinical investigation, non-interventional and non-randomized. The overall goal of this clinical study is to generate additional clinical data confirming the safety and efficacy of the remote programming functionality of Target CI version 1.5 and the AB Remote Support app. Hearing outcomes are expected to be similar whether a study subject's sound processor is programmed in the traditional method in the audiologist's office or whether programming is performed via remote fitting. Therefore, the study uses a non-inferiority design to determine whether sentence recognition in noise is no worse with remote fitting than in an in-office setting.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Ability to give feedback on hearing impressions
* Aged 18 years of age or older
* Implanted with a HiResolution Bionic Ear System (HiRes 90K or HiRes 90K Advantage or HiRes Ultra or HiRes Ultra 3D) on at least one side

  * Group 1 - Unilateral: no hearing device except contralateral routing of signals (CROS) device on the contralateral side
  * Group 2 - Bilateral: implanted on both sides
  * Group 3 - Bimodal: hearing aid on the contralateral side
* Minimum of six months of cochlear implant experience
* Minimum of one month experience with a Naída CI M or Sky CI M sound processor
* Fluent in French language
* Ability to be tested via speech perception test in noise
* Smartphone user

Exclusion Criteria:

* Clinical presentation indicative of potential implanted device malfunction
* Unrealistic expectations regarding potential benefits, risks and limitations of the investigational device as determined by the Investigator
* Unwillingness or inability of subject to comply with all investigational requirements as determined by the Investigator

Pregnancy and breast-feeding are not exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced Bionics adults CI users
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
50% SRT measured as signal to noise ratio in DB (French Matrix test in noise) | one-month chronic use of remotely fitted sound processor
  The primary efficacy objective is to demonstrate that speech recognition in noise after remote fitting is no worse than speech recognition in noise after in-office fitting.

SECONDARY OUTCOMES:
Score in the Lafon phoneme test in quiet | one-month chronic use of remotely fitted sound processor
  The secondary efficacy objective is to demonstrate that speech recognition in quiet after remote fitting is no worse than speech recognition in quiet after in-office fitting.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupement Hospitalier Pitié Salpêtrière, Paris, France